CLINICAL TRIAL: NCT01008475
Title: An Open-label, Randomized, Controlled, Multicenter, Phase I/II Trial Investigating 2 EMD 525797 Doses in Combination With Cetuximab and Irinotecan Versus Cetuximab and Irinotecan Alone, as Second-line Treatment for Subjects With K-ras Wild Type Metastatic Colorectal Cancer (mCRC)
Brief Title: EMD 525797 in Combination With Cetuximab and Irinotecan in K-ras Wild Type Metastatic Colorectal Cancer
Acronym: POSEIDON
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EMR62242-004
Record Dates: First submitted 2009-10-19; First posted 2009-11-05 (Estimated); Results first posted 2016-03-30 (Estimated); Last update posted 2016-03-30 (Estimated); Status verified 2016-02

CONDITIONS: Metastatic Colorectal Cancer
Keywords: EMD 525797; Cetuximab; Irinotecan; metastatic colorectal cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Abituzumab; Cetuximab; Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (7):
- Safety part: EMD 525797 250 mg + Standard of Care (SoC) (Experimental): EMD 525797 250 mg in combination with cetuximab and irinotecan
  Interventions: Drug: EMD 525797 250 mg; Drug: Cetuximab; Drug: Irinotecan
- Safety part: EMD 525797 500 mg + SoC (Experimental): EMD 525797 500 mg in combination with cetuximab and irinotecan
  Interventions: Drug: EMD 525797 500 mg; Drug: Cetuximab; Drug: Irinotecan
- Safety part: EMD 525797 750 mg + SoC (Experimental): EMD 525797 750 mg in combination with cetuximab and irinotecan
  Interventions: Drug: EMD 525797 750 mg; Drug: Cetuximab; Drug: Irinotecan
- Safety part: EMD 525797 1000 mg + SoC (Experimental): EMD 525797 1000 mg in combination with cetuximab and irinotecan
  Interventions: Drug: EMD 525797 1000 mg; Drug: Cetuximab; Drug: Irinotecan
- Randomized part: EMD 525797 500 mg + SoC (Experimental): EMD 525797 500 mg in combination with cetuximab and irinotecan
  Interventions: Drug: EMD 525797 500 mg; Drug: Cetuximab; Drug: Irinotecan
- Randomized Part: EMD 525797 1000 mg + SoC (Experimental): EMD 525797 1000 mg (or dose as defined by safety monitoring committee (SMC)] in combination with cetuximab and irinotecan.
  Interventions: Drug: EMD 525797 1000 mg; Drug: Cetuximab; Drug: Irinotecan
- Randomized Part: SoC (Other): Cetuximab and irinotecan
  Interventions: Drug: Cetuximab; Drug: Irinotecan

INTERVENTIONS:
Drug: EMD 525797 250 mg — EMD 525797 will be administered at a target dose of 250 mg as a 1-hour intravenous infusion for every 2 week until radio-graphically documented PD (as assessed by the investigator), unacceptable toxicity or eligibility for curative resection (investigator's assessment), or withdrawal of consent .
  Arms: Safety part: EMD 525797 250 mg + Standard of Care (SoC)
Drug: EMD 525797 500 mg — Safety part: EMD 525797 will be administered at a target dose of 500 mg as a 1-hour intravenous infusion for every 2 weeks until radio-graphically documented PD (as assessed by the investigator), unacceptable toxicity or eligibility for curative resection (investigator's assessment), or withdrawal of consent .
  Randomized part: EMD 525797 will be administered at a target dose of 500 mg as a 1-hour intravenous infusion for every 2 weeks until radio-graphically documented PD (as assessed by the investigator), unacceptable toxicity or eligibility for curative resection (investigator's assessment), or withdrawal of consent.
  Arms: Randomized part: EMD 525797 500 mg + SoC; Safety part: EMD 525797 500 mg + SoC
Drug: EMD 525797 750 mg — EMD 525797 will be administered at a target dose of 750 mg as a 1-hour intravenous infusion for every 2 weeks until radio-graphically documented PD (as assessed by the investigator), unacceptable toxicity or eligibility for curative resection (investigator's assessment), or withdrawal of consent .
  Other Names: Abituzumab
  Arms: Safety part: EMD 525797 750 mg + SoC
Drug: EMD 525797 1000 mg — Safety part: EMD 525797 will be administered at a target dose of 1000 mg as a 1-hour intravenous infusion for every 2 weeks until radio-graphically documented PD (as assessed by the investigator), unacceptable toxicity or eligibility for curative resection (investigator's assessment), or withdrawal of consent .
  Randomized part: EMD 525797 will be administered at a target dose of 1000 mg as a 1-hour intravenous infusion for every 2 weeks until radio-graphically documented PD (as assessed by the investigator), unacceptable toxicity or eligibility for curative resection (investigator's assessment), or withdrawal of consent.
  Other Names: Abituzumab
  Arms: Randomized Part: EMD 525797 1000 mg + SoC; Safety part: EMD 525797 1000 mg + SoC
Drug: Cetuximab — Safety part: Cetuximab will be administered at a dose of 400 milligram per square meter (mg/m^2) on Day 1 Cycle 1 (Week 1) as IV infusion for 2 hours, and then at a dose of 250 mg/m^2 on Day 8 (Week 2) once weekly until DLT.
  Randomized part: Cetuximab will be administered at a dose of 400 milligram per square meter (mg/m^2) on Day 1 Cycle 1 (Week 1) as IV infusion for 2 hours, and then at a dose of 250 mg/m^2 on Day 8 (Week 2) once weekly until radio-graphically documented PD (as assessed by the investigator), unacceptable toxicity or eligibility for curative resection (investigator's assessment), or withdrawal of consent.
Drug: Irinotecan — Safety part: Irinotecan will be administered at a dose of 180 mg/m^2 as IV infusion for 30-90 minutes for every 2 weeks until radio-graphically documented PD (as assessed by the investigator), unacceptable toxicity or eligibility for curative resection (investigator's assessment), or withdrawal of consent .
  Randomized part: Irinotecan will be administered at a dose of 180 mg/m^2 as IV infusion for 30-90 minutes for every 2 weeks until radio-graphically documented PD (as assessed by the investigator), unacceptable toxicity or eligibility for curative resection (investigator's assessment), or withdrawal of consent.

SUMMARY:
The purpose of this study is to assess the safety and clinical activity of the experimental drug EMD 525797 (study drug), a monoclonal antibody targeting alfa integrins, in combination with irinotecan and cetuximab in K-ras wildtype metastatic colorectal cancer patients.

ELIGIBILITY:
Inclusion Criteria:

Subjects with histologically confirmed kras wildtype (WT) colorectal carcinoma (CRC) with documented distant metastasis

* Prior oxaliplatin/fluoropyrimidine-containing regimen for the first-line treatment of metastatic disease
* Failed an oxaliplatin regimen for metastatic colorectal carcinoma (mCRC). Failure is defined as either progressive disease (PD) (clinical or radiologic) within 6 months of the last dose of any agent of an oxaliplatin-based regimen or intolerance to an oxaliplatin regimen. Intolerance to an oxaliplatin regimen is defined as discontinuation due to any of the following: severe allergic reaction, persistent severe neurotoxicity, or delayed recovery from toxicity preventing retreatment
* At least 1 radiographically documented measurable lesion in a previously non irradiated area according to Response Evaluation Criteria In Solid Tumors (RECIST, Version 1.0), i.e., this lesion must be adequately measurable in at least 1 dimension (longest diameter to be recorded) as greater than or equal to (>=) 2 centimeter (cm) by conventional techniques or >=1 cm by spiral computed tomography (CT) scan
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1, or Karnofsky performance status (KPS) >= 80 percent (%)
* Absolute Neutrophil Count (ANC) >=1.5 x 10^9/Liter
* Platelets >=100 x 10^9/Liter
* Hemoglobin >=9 gram per deciliter (g/dL) (without transfusions)
* Bilirubin less than or equal to (<=) 1.5 x upper limit normal (ULN)
* Aspartate transaminase (AST) <=5 x ULN and alanine transaminase (ALT) <=5 x ULN
* Serum creatinine <=1.25 x ULN and/or creatinine clearance >=50 milliliter per minute (mL/min)
* International Nationalized Ratio (INR), and partial thromboplastin time (PTT) within normal limits
* Sodium and potassium within normal limits or <=10% above or below (supplementation permitted)

Exclusion Criteria:

* Previous treatment with any inhibitor of Epidermal Growth Factor Receptor (EGFR)
* Known brain metastasis and/or leptomeningeal disease
* Radiotherapy (except localized radiotherapy for pain relief), major surgery, or any investigational drug in the 30 days before the start of trial treatment entry; planned major surgery during the trial
* Concurrent chronic systemic immune or hormone therapy not indicated in this trial protocol (except for physiologic replacement; steroids up to 10 mg of prednisone equivalent or topical and inhaled steroids are allowed)
* Clinically relevant coronary artery disease (New York Heart Association [NYHA] functional angina classification III/IV), congestive heart failure (NYHA III/IV), clinically relevant cardiomyopathy, history of myocardial infarction in the last 12 months, or high risk of uncontrolled arrhythmia
* Uncontrolled hypertension defined as systolic blood pressure >=160 millimeter of mercury (mmHg) and/or diastolic blood pressure >=100 mmHg under resting conditions
* History of coagulation disorder associated with bleeding or recurrent thrombotic events
* History of recent peptic ulcer disease (endoscopically proven gastric, duodenal or esophageal ulcer) within 6 months of trial treatment start
* Chronic inflammatory bowel disease, or acute/chronic ileus
* Active infection (requiring i.v. antibiotics), including active tuberculosis, active or chronic Hepatitis B or C, or ongoing HIV infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 232 (Actual)
Dates: Start 2009-10; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — Merck KGaA, Darmstadt, Germany; Prof. Josep Tabernero, Principal Investigator — HU Vall d' Hebron, Servei d'oncologia. E difici General
Locations (62):
- Belgium (4):
  - Research Site, Brussels
  - Research Site, Edegem
  - Research Site, Ghent
  - Research Site, Leuven
- Research Site, Sofia, Bulgaria
- Research Site, Stróvolos, Nicosia, Cyprus
- Czechia (6):
  - Research Site, Brno
  - Research Site, Hořovice
  - Research Site, Kutná Hora
  - Research Site, Olomouc
  - Research Site, Pardubice
  - Research Site, Prague
- Germany (11):
  - Research Site, Dresden
  - Research Site, Essen
  - Research Site, Freiburg im Breisgau
  - Research Site, Hamburg
  - Research site, Hanover
  - Research Site, Heilbronn
  - Research Site, Landshut
  - Research Site, Leipzig
  - Research Site, Munich
  - Research Site, Recklinghausen
  - Research Site, Ulm
- Greece (2):
  - Research Site, Thessaloniki, Cyprus
  - Research Site, Mournies Chania
- Hungary (6):
  - Research Site, Budapest
  - Research Site, Győr
  - Research Site, Kecskemét
  - Research Site, Miskolc
  - Research Site, Nyíregyháza
  - Research Site, Szolnok
- Israel (5):
  - Research Site, Haifa
  - Research Site, Jerusalem
  - Research Site, Ramat Gan
  - Research Site, Rehovot
  - Research Site, Tel Aviv
- Poland (6):
  - Research Site, Elblag
  - Research Site, Gdansk
  - Research Site, Gliwice
  - Research Site, Lodz
  - Research Site, Rybnik
  - Research Site, Warsaw
- Russia (6):
  - Research, Arkhangelsk
  - Research Site, Moscow
  - Research Site, Novosibirsk
  - Research Site, Omsk
  - Research Site, Saint Petersburg
  - Research Site, Tomsk
- Spain (8):
  - Research Site, Barcelona
  - Research Site, Elche
  - Research Site, Madrid
  - Research Site, Mallorca
  - Research Site, Santander
  - Research Site, Santiago de Compostela
  - Research Site, Terrassa
  - Research Site, Valencia
- United Kingdom (6):
  - Research Site, Aberdeen
  - Research Site, Glasgow
  - Research Site, London
  - Research Site, Manchester
  - Research Site, Nottingham
  - Research Site, Sutton

REFERENCES:
- [Derived] Elez E, Kocakova I, Hohler T, Martens UM, Bokemeyer C, Van Cutsem E, Melichar B, Smakal M, Csoszi T, Topuzov E, Orlova R, Tjulandin S, Rivera F, Straub J, Bruns R, Quaratino S, Tabernero J. Abituzumab combined with cetuximab plus irinotecan versus cetuximab plus irinotecan alone for patients with KRAS wild-type metastatic colorectal cancer: the randomised phase I/II POSEIDON trial. Ann Oncol. 2015 Jan;26(1):132-140. doi: 10.1093/annonc/mdu474. Epub 2014 Oct 15. PMID 25319061

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This study consists of two parts, safety part and randomized part. A total of 16 subjects were included in the safety part and 216 subjects were included in the randomized part of the study. The subjects who participated in the safety part of the study were not included in the randomized part of the study.
Groups:
- Safety Part: EMD 525797 250 mg + SoC: Cetuximab was administered at a dose of 400 mg/m^2 on Day 1 Cycle 1 (Week 1) as IV infusion for 2 hours, and then at a dose of 250 mg/m^2 on Day 8 (Week 2) once weekly; followed by EMD 525797 at a target dose of 250 mg as a 1-hour IV infusion for every 2 weeks, followed by Irinotecan at a dose of 180 mg/m^2 as IV infusion for 30-90 minutes for every 2 weeks until radio-graphically documented progressive disease (PD) (as assessed by the investigator), unacceptable toxicity or eligibility for curative resection (investigator's assessment), or withdrawal of consent.
- Safety Part: EMD 525797 500 mg + SoC; Randomized Part: EMD 525797 500 mg + SoC: Cetuximab was administered at a dose of 400 mg/m^2 on Day 1 Cycle 1 (Week 1) as IV infusion for 2 hours, and then at a dose of 250 mg/m^2 on Day 8 (Week 2) once weekly; followed by EMD 525797 at a target dose of 500 mg as a 1-hour IV infusion for every 2 weeks, followed by Irinotecan at a dose of 180 mg/m^2 as IV infusion for 30-90 minutes for every 2 weeks until radio-graphically documented progressive disease (PD) (as assessed by the investigator), unacceptable toxicity or eligibility for curative resection (investigator's assessment), or withdrawal of consent.
- Safety Part: EMD525797 750 mg + SoC: Cetuximab was administered at a dose of 400 mg/m^2 on Day 1 Cycle 1 (Week 1) as IV infusion for 2 hours, and then at a dose of 250 mg/m^2 on Day 8 (Week 2) once weekly; followed by EMD 525797 at a target dose of 750 mg as a 1-hour IV infusion for every 2 weeks, followed by Irinotecan at a dose of 180 mg/m^2 as IV infusion for 30-90 minutes for every 2 weeks until radio-graphically documented progressive disease (PD) (as assessed by the investigator), unacceptable toxicity or eligibility for curative resection (investigator's assessment), or withdrawal of consent.
- Safety Part: EMD 525797 1000 mg +SoC; Randomized Part: EMD 525797 1000 mg + SoC: Cetuximab was administered at a dose of 400 mg/m^2 on Day 1 Cycle 1 (Week 1) as IV infusion for 2 hours, and then at a dose of 250 mg/m^2 on Day 8 (Week 2) once weekly; followed by EMD 525797 at a target dose of 1000 mg as a 1-hour IV infusion for every 2 weeks, followed by Irinotecan at a dose of 180 mg/m^2 as IV infusion for 30-90 minutes for every 2 weeks until radio-graphically documented progressive disease (PD) (as assessed by the investigator), unacceptable toxicity or eligibility for curative resection (investigator's assessment), or withdrawal of consent.
- Randomized Part: Standard of Care (SoC): Cetuximab was administered at a dose of 400 milligram per square meter (mg/m^2) on Day 1 Cycle 1 (Week 1) as intravenous (IV) infusion for 2 hours, and then at a dose of 250 mg/m^2 on Day 8 (Week 2) once weekly followed by irinotecan at a dose of 180 mg/m^2 as IV infusion for 30-90 minutes for every 2 weeks until radio-graphically documented progressive disease (PD) (as assessed by the investigator), unacceptable toxicity or eligibility for curative resection (investigator's assessment), or withdrawal of consent.
Period: Overall Study
Arm/Group | Safety Part: EMD 525797 250 mg + SoC | Safety Part: EMD 525797 500 mg + SoC | Safety Part: EMD525797 750 mg + SoC | Safety Part: EMD 525797 1000 mg +SoC | Randomized Part: Standard of Care (SoC) | Randomized Part: EMD 525797 500 mg + SoC | Randomized Part: EMD 525797 1000 mg + SoC
Started | 3 | 3 | 7 | 3 | 72 | 73 | 71
Safety Analysis Set | 3 | 3 | 7 | 3 | 73 (1 subject randomized to EMD525797 1000 mg group received only SoC. Hence, reported under SOC group.) | 72 | 69
Completed | 3 | 3 | 7 | 3 | 67 | 67 | 67
Not Completed | 0 | 0 | 0 | 0 | 5 | 6 | 4
Not completed — Ongoing treatment at data cut-off date | 0 | 0 | 0 | 0 | 5 | 6 | 4

BASELINE CHARACTERISTICS:
Population: All the subjects who were enrolled in to the study (safety and randomized part).
Groups:
- Safety Part: EMD 525797 250 mg + Standard of Care (SoC): Cetuximab was administered at a dose of 400 milligram per square meter (mg/m^2) on Day 1 as IV infusion for 2 hours, and then at a dose of 250 mg/m^2 on Day 8 once weekly followed by EMD 525797 at a target dose of 250 mg as a 1-hour IV infusion for every 2 weeks, followed by irinotecan at a dose of 180 mg/m^2 as IV infusion for 30-90 minutes for every 2 weeks until radio-graphically documented progressive disease (PD) (as assessed by the investigator), unacceptable toxicity or eligibility for curative resection (investigator's assessment), or withdrawal of consent.
- Safety Part: EMD 525797 500 mg + SoC: Cetuximab was administered at a dose of 400 milligram per square meter (mg/m^2) on Day 1 as IV infusion for 2 hours, and then at a dose of 250 mg/m^2 on Day 8 once weekly followed by EMD 525797 at a target dose of 500 mg as a 1-hour IV infusion for every 2 weeks, followed by irinotecan at a dose of 180 mg/m^2 as IV infusion for 30-90 minutes for every 2 weeks until radio-graphically documented progressive disease (PD) (as assessed by the investigator), unacceptable toxicity or eligibility for curative resection (investigator's assessment), or withdrawal of consent.
- Safety Part: EMD 525797 750 mg + SoC: Cetuximab was administered at a dose of 400 milligram per square meter (mg/m^2) on Day 1 as IV infusion for 2 hours, and then at a dose of 250 mg/m^2 on Day 8 once weekly followed by EMD 525797 at a target dose of 750 mg as a 1-hour IV infusion for every 2 weeks, followed by irinotecan at a dose of 180 mg/m^2 as IV infusion for 30-90 minutes for every 2 weeks until radio-graphically documented progressive disease (PD) (as assessed by the investigator), unacceptable toxicity or eligibility for curative resection (investigator's assessment), or withdrawal of consent.
- Safety Part: EMD 525797 1000 mg + SoC: Cetuximab was administered at a dose of 400 milligram per square meter (mg/m^2) on Day 1 as IV infusion for 2 hours, and then at a dose of 250 mg/m^2 on Day 8 once weekly followed by EMD 525797 at a target dose of 1000 mg as a 1-hour IV infusion for every 2 weeks, followed by irinotecan at a dose of 180 mg/m^2 as IV infusion for 30-90 minutes for every 2 weeks until radio-graphically documented progressive disease (PD) (as assessed by the investigator), unacceptable toxicity or eligibility for curative resection (investigator's assessment), or withdrawal of consent.
- Randomized Part: SoC: Cetuximab was administered at a dose of 400 milligram per square meter (mg/m^2) on Day 1 Cycle 1 (Week 1) as intravenous (IV) infusion for 2 hours, and then at a dose of 250 mg/m^2 on Day 8 (Week 2) once weekly followed by irinotecan at a dose of 180 mg/m^2 as IV infusion for 30-90 minutes for every 2 weeks until radio-graphically documented progressive disease (PD) (as assessed by the investigator), unacceptable toxicity or eligibility for curative resection (investigator's assessment), or withdrawal of consent.
- Total: Total of all reporting groups
Arm/Group | Safety Part: EMD 525797 250 mg + Standard of Care (SoC) | Safety Part: EMD 525797 500 mg + SoC | Safety Part: EMD 525797 750 mg + SoC | Safety Part: EMD 525797 1000 mg + SoC | Randomized Part: SoC | Randomized Part: EMD 525797 500 mg + SoC | Randomized Part: EMD 525797 1000 mg + SoC | Total
Number analyzed (Participants) | 3 | 3 | 7 | 3 | 72 | 73 | 71 | 232
Age, Continuous [Mean (Standard Deviation); unit: Years] | 62.3 (11.5) | 57.7 (11.2) | 60.4 (6.2) | 63.0 (7.2) | 56.2 (12.11) | 58.9 (12.18) | 59.9 (10.63) | 58.5 (11.49)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 4 | 2 | 27 | 36 | 23 | 95
  Male | 1 | 2 | 3 | 1 | 45 | 37 | 48 | 137

OUTCOME MEASURES:

1. Primary Outcome: Safety Part: Number of Subjects Experiencing DLTs (Dose Limiting Toxicity)
Description: DLT was defined as any Grade 4 hematologic toxicity or Grade 3/4 non-hematologic toxicity assessed as related to trial treatment by the Investigator and/or Sponsor and confirmed by the safety monitoring committee (SMC) to be relevant to the combination treatment within the first cycle of therapy. Any Grade 3 or 4 non haematological toxicity, any Grade 4 hematological toxicity, treatment related deaths within the first 2 weeks of therapy. Toxicities excluded from DLT: alopecia, rash, nausea, vomiting and hypomagnesemia of Grade 3 or 4 severity, Grade 4 neutropenia or leukopenia lasting for =< 5 days and not associated with fever; Single laboratory values out of normal range without any clinical correlation and resolve within 7 days; Grade 3 or 4 diarrhoea without adequate supportive care. Adequate supportive care has been administered and Grade 4 diarrhea persists (investigator decision); isolated Grade 4 lymphocytopenia and thrombocytopenia without clinical correlation.
Time Frame: Time from the first dose of study drug up to 2 weeks
Population: Dose-escalation analysis set included subjects who received atleast 1 dose of EMD 525797 and who met atleast 1 of the following: Did not withdraw before the end of DLT evaluation period (2 weeks from 1st drug intake) for reasons other than DLT;those who experienced a DLT during this period and received 1 dose of EMD 525797 as per cohort allocation.
Measure: Number; unit: subjects
Arm/Group | Safety Part: EMD 525797 250 mg + SoC | Safety Part: EMD 525797 500 mg + SoC | Safety Part: EMD525797 750 mg + SoC | Safety Part: EMD 525797 1000 mg +SoC
Number analyzed (Participants) | 3 | 3 | 7 | 3
subjects | 0 | 0 | 0 | 0

2. Primary Outcome: Randomized Part: Progression Free Survival (PFS)
Description: PFS was defined as the time from the randomization date to first documented sign of objective radio-graphic disease progression (PD) as per Response Evaluation Criteria In Solid Tumors version 1. (RECIST 1.0) or death from any cause if reported within 12 weeks from the last tumor assessment. PD per RECIST v 1.0 was defined as at least 20% increase in the sum of the longest diameter of target lesions, taking as the reference the smallest sum of longest diameters recorded since treatment started, or unequivocal progression of existing non-target lesion or appearance of new lesions. Subjects who did not progress or died at the time of analyses, or subjects who died without previously radio-graphically documented PD and death was observed after more than 12 weeks of last tumor assessment without progression, these subjects were censored at their last tumor assessment date or date of randomization, whichever occurred last.
Time Frame: Time from randomization until progressive disease or death; assessed up to 18 months (i.e data cut-off date: 09 Oct 2013)
Population: Intention-to-treat (ITT) analysis set included all the subjects who were randomized into the treatment groups.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Standard of Care (SoC): Cetuximab was administered at a dose of 400 milligram per square meter (mg/m^2) on Day 1 Cycle 1 (Week 1) as intravenous (IV) infusion for 2 hours, and then at a dose of 250 mg/m^2 on Day 8 (Week 2) once weekly followed by irinotecan at a dose of 180 mg/m^2 as IV infusion for 30-90 minutes for every 2 weeks until radiographically documented progressive disease (PD) (as assessed by the investigator), unacceptable toxicity or eligibility for curative resection (investigator's assessment), or withdrawal of consent.
- EMD 525797 500 mg + SoC: Cetuximab was administered at a dose of 400 mg/m^2 on Day 1 Cycle 1 (Week 1) as IV infusion for 2 hours, and then at a dose of 250 mg/m^2 on Day 8 (Week 2) once weekly; followed by EMD 525797 at a target dose of 500 mg as a 1-hour IV infusion for every 2 weeks, followed by Irinotecan at a dose of 180 mg/m^2 as IV infusion for 30-90 minutes for every 2 weeks until radiographically documented PD (as assessed by the investigator), unacceptable toxicity or eligibility for curative resection (investigator's assessment), or withdrawal of consent.
- EMD 525797 1000 mg + SoC: Cetuximab was administered at a dose of 400 mg/m^2 on Day 1 Cycle 1 (Week 1) as IV infusion for 2 hours, and then at a dose of 250 mg/m^2 on Day 8 (Week 2) once weekly; followed by EMD 525797 at a target dose of 1000 mg as a 1-hour IV infusion for every 2 weeks, followed by Irinotecan at a dose of 180 mg/m^2 as IV infusion for 30-90 minutes for every 2 weeks until radio-graphically documented progressive disease (PD) (as assessed by the investigator), unacceptable toxicity or eligibility for curative resection (investigator's assessment), or withdrawal of consent.
Arm/Group | Standard of Care (SoC) | EMD 525797 500 mg + SoC | EMD 525797 1000 mg + SoC
Number analyzed (Participants) | 72 | 73 | 71
months | 5.6 [4.2 to 6.9] | 5.4 [4.1 to 6.0] | 5.6 [4.1 to 6.9]
Statistical Analysis 1: Comparison: Standard of Care (SoC) vs EMD 525797 500 mg + SoC; Test type: Superiority or Other; Cox Proportional Hazard = 1.13, 95% CI 2-sided [0.78 to 1.64]
Statistical Analysis 2: Comparison: Standard of Care (SoC) vs EMD 525797 1000 mg + SoC; Test type: Superiority or Other; Cox Proportional Hazard = 1.11, 95% CI 2-sided [0.77 to 1.61]

3. Secondary Outcome: Overall Survival (OS) Time
Description: OS was defined as the time from the date of randomization to the date of death from any cause. For subjects who were still alive at the analysis cut off date or lost to follow up, survival was censored at the last recorded date the subject was known to be alive or at the analysis cut off date, whichever occurred first.
Time Frame: Time from randomization until death assessed up to 18 months (i.e data cut-off date: 09 Oct 2013)
Population: ITT analysis set included all the subjects who were randomized into the trial.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Standard of Care (SoC) | EMD 525797 500 mg + SoC | EMD 525797 1000 mg + SoC
Number analyzed (Participants) | 72 | 73 | 71
months | 11.6 [9.8 to 15.7] | 15.0 [10.9 to 19.2] | 14.4 [9.8 to 19.3]
Statistical Analysis 1: Comparison: Standard of Care (SoC) vs EMD 525797 500 mg + SoC; Test type: Superiority or Other; Cox Proportional Hazard = 0.83, 95% CI 2-sided [0.54 to 1.28]
Statistical Analysis 2: Comparison: Standard of Care (SoC) vs EMD 525797 1000 mg + SoC; Test type: Superiority or Other; Cox Proportional Hazard = 0.80, 95% CI 2-sided [0.52 to 1.25]

4. Secondary Outcome: Time to Progression (TTP)
Description: TTP was defined as the time from the date of randomization to the date of objective radiographic disease progression (PD). PD per RECIST v 1.0 was defined as at least 20% increase in the sum of the longest diameter of target lesions, taking as the reference the smallest sum of longest diameters recorded since treatment started, or unequivocal progression of existing non-target lesion or appearance of new lesions. For subjects who did not progress or who were without any post baseline tumor assessment, TTP was censored at their last tumor assessment date, or at the randomization date, whichever occurred last.
Time Frame: Time from randomization until disease progression assessed up to 18 months (i.e data cut-off date: 09 Oct 2013)
Population: ITT analysis set included all the subjects who were randomized into the trial.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Standard of Care (SoC) | EMD 525797 500 mg + SoC | EMD 525797 1000 mg + SoC
Number analyzed (Participants) | 72 | 73 | 71
months | 5.8 [4.4 to 7.2] | 5.6 [4.2 to 8.3] | 6.5 [4.2 to 7.1]
Statistical Analysis 1: Comparison: Standard of Care (SoC) vs EMD 525797 500 mg + SoC; Test type: Superiority or Other; Cox Proportional Hazard = 1.11, 95% CI 2-sided [0.75 to 1.65]
Statistical Analysis 2: Comparison: Standard of Care (SoC) vs EMD 525797 1000 mg + SoC; Test type: Superiority or Other; Cox Proportional Hazard = 1.11, 95% CI 2-sided [0.75 to 1.65]

5. Secondary Outcome: Number of Subjects With Tumor Response
Description: Tumor response was defined as the presence of at least 1 confirmed complete response (CR) or confirmed partial response (PR) as judged by RECIST version 1.0. CR was defined for target lesions (TLs) as the disappearance of all lesions, and for non-target lesions (NTLs) as the disappearance of all non-target non-measurable lesions and/or normalization of serum levels of tumor markers. PR was defined for TLs as at least a 30 percent (%) decrease from baseline (BL) in the sum of longest diameter (SLD) of TLs.
Time Frame: Time from randomization up to 18 months (i.e data cut-off date: 09 Oct 2013)
Population: ITT analysis set included all the subjects who were randomized into the trial.
Measure: Number; unit: Subjects
Arm/Group | Standard of Care (SoC) | EMD 525797 500 mg + SoC | EMD 525797 1000 mg + SoC
Number analyzed (Participants) | 72 | 73 | 71
Subjects
  CR | 2 | 1 | 0
  PR | 17 | 19 | 18

6. Secondary Outcome: Time to Treatment Failure (TTF)
Description: TTF was defined as the time from randomization to treatment discontinuation for any reason. For subjects on drug at the analysis cut off date or lost to follow up, TTF was censored at the trial discontinuation date or at the analysis cut off date, whichever occurred first.
Time Frame: Time from randomization until discontinuation assessed up to 18 months (i.e data cut-off date: 09 Oct 2013)
Population: ITT analysis set included all the subjects who were randomized into the trial.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Standard of Care (SoC) | EMD 525797 500 mg + SoC | EMD 525797 1000 mg + SoC
Number analyzed (Participants) | 72 | 73 | 71
months | 5.2 [4.4 to 6.2] | 4.3 [3.6 to 6.1] | 4.8 [3.3 to 6.6]
Statistical Analysis 1: Comparison: Standard of Care (SoC) vs EMD 525797 500 mg + SoC; Test type: Superiority or Other; Cox Proportional Hazard = 0.95, 95% CI 2-sided [0.67 to 1.34]
Statistical Analysis 2: Comparison: Standard of Care (SoC) vs EMD 525797 1000 mg + SoC; Test type: Superiority or Other; Cox Proportional Hazard = 1.05, 95% CI 2-sided [0.74 to 1.48]

ADVERSE EVENTS:
Time Frame: From the first dose of study drug administration up to 50 days after the last dose of study drug administration
Description: The safety analysis set included all subjects who received at least 1 dose of the trial medication. 1 subject who was randomized to EMD525797 1000 mg group received only SoC, therefore this subjects was reported under the SOC group.
Arm/Group | Safety Part: EMD 525797 250 mg + SoC | Safety Part: EMD 525797 500 mg + SoC | Safety Part: EMD525797 750 mg + SoC | Safety Part: EMD 525797 1000 mg +SoC | Standard of Care (SoC) | EMD 525797 500 mg + SoC | EMD 525797 1000 mg + SoC
Serious Adverse Events (participants affected / at risk) | 2/3 | 2/3 | 3/7 | 3/3 | 30/73 | 27/72 | 34/69
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 7/7 | 3/3 | 72/73 | 72/72 | 68/69
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Safety Part: EMD 525797 250 mg + SoC (N=3) | Safety Part: EMD 525797 500 mg + SoC (N=3) | Safety Part: EMD525797 750 mg + SoC (N=7) | Safety Part: EMD 525797 1000 mg +SoC (N=3) | Standard of Care (SoC) (N=73) | EMD 525797 500 mg + SoC (N=72) | EMD 525797 1000 mg + SoC (N=69)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Febrile Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 3 (3) | 3 (4)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 3 (3)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Atrial Fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Cardiac Failure Acute (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tachyarrhythmia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Inappropriate Antidiuretic Hormone Secretion (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal Hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 5 (5)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Colonic Obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 7 (7)
Enteritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Enterovesical Fistula (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal Stenosis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal Toxicity (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (3) | 0 (0)
Gastrointestinal Ulcer Haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Intestinal Obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Intestinal Perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (2)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (3) | 2 (2)
Periodontitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Subileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 2 (4) | 2 (2)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 1 (1)
Death (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Device Malfunction (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Disease Progression (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 2 (3) | 3 (4)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
General Physical Health Deterioration (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Mucosal Inflammation (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Multi-Organ Failure (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Performance Status Decreased (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hepatic Failure (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Jaundice Cholestatic (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anaphylactic Shock (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal Wall Abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Device Related Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Device Related Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Erysipelas (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Febrile Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Peritonitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Rectal Abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 1 (2)
Septic Shock (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Femoral Neck Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Overdose (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Blood Bilirubin Increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood Creatinine Increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Coagulation Factor Increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gamma-Glutamyltransferase Increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
General Physical Condition Abnormal (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutrophil Count Decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cachexia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Decreased Appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 2 (2)
Diabetes Mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Electrolyte Imbalance (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neck Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pathological Fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cerebrovascular Accident (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Coma (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Epilepsy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Polyneuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Renal Failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Renal Failure Acute (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea Exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (5) | 0 (0) | 2 (2)
Respiratory Disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Toxic Skin Eruption (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Thrombosis Prophylaxis (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Deep Vein Thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Venous Thrombosis Limb (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Safety Part: EMD 525797 250 mg + SoC (N=3) | Safety Part: EMD 525797 500 mg + SoC (N=3) | Safety Part: EMD525797 750 mg + SoC (N=7) | Safety Part: EMD 525797 1000 mg +SoC (N=3) | Standard of Care (SoC) (N=73) | EMD 525797 500 mg + SoC (N=72) | EMD 525797 1000 mg + SoC (N=69)
Agranulocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 1 (3) | 0 (0) | 0 (0) | 1 (1) | 9 (28) | 15 (40) | 18 (33)
Anaemia Of Malignant Disease (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (7) | 0 (0)
Aplastic Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (6) | 1 (3)
Granulocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0)
Haemorrhagic Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypochromic Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Iron Deficiency Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (5) | 2 (8) | 1 (5)
Leukocytosis (Blood and lymphatic system disorders) | 1 (9) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 3 (3) | 4 (5)
Leukopenia (Blood and lymphatic system disorders) | 2 (3) | 1 (1) | 3 (6) | 2 (4) | 14 (63) | 14 (55) | 16 (70)
Lymphadenitis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Microcytic Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Neutropenia (Blood and lymphatic system disorders) | 1 (3) | 0 (0) | 1 (1) | 2 (5) | 24 (96) | 26 (91) | 26 (85)
Normochromic Normocytic Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Splenic Vein Thrombosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 7 (17) | 2 (3) | 3 (4)
Thrombocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Angina Pectoris (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Atrial Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Left Ventricular Dysfunction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Myocardial Ischaemia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Right Ventricular Dysfunction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sinus Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
Supraventricular Extrasystoles (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Ventricular Extrasystoles (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Congenital Hair Disorder (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Trichomegaly (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
External Ear Inflammation (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypoacusis (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Vertigo Positional (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypothyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 0 (0)
Blepharitis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (2)
Conjunctivitis (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 9 (21) | 4 (6) | 8 (14)
Dry Eye (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Erythema Of Eyelid (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eye Pain (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eyelid Oedema (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Eyelid Pain (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eyelids Pruritus (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Iritis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Meibomianitis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Miosis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ocular Hyperaemia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ocular Icterus (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vision Blurred (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Visual Acuity Reduced (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Visual Impairment (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Abdominal Discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Abdominal Distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 2 (2) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 11 (18) | 14 (24) | 18 (24)
Abdominal Pain Lower (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Abdominal Pain Upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (8) | 5 (5) | 6 (7)
Abdominal Tenderness (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anal Haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Anorectal Discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Aphthous Stomatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 2 (2) | 4 (4) | 9 (16)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 3 (3) | 0 (0)
Cheilitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 7 (14) | 7 (13) | 15 (22)
Diarrhoea (Gastrointestinal disorders) | 1 (2) | 0 (0) | 4 (10) | 2 (15) | 31 (128) | 48 (197) | 45 (209)
Dry Mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (2)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 4 (6) | 5 (6) | 2 (2)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Enteritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Enterovesical Fistula (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Faecal Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 7 (8)
Food Poisoning (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Frequent Bowel Movements (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastritis Erosive (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal Disorder (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (3)
Gastrointestinal Motility Disorder (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal Toxicity (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
Gastrooesophageal Sphincter Insufficiency (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gingival Bleeding (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haemorrhoidal Haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 3 (3) | 2 (2)
Intestinal Fistula (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Intestinal Haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intestinal Villi Atrophy (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lip Ulceration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mesenteric Vein Thrombosis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mouth Ulceration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 1 (2)
Mucous Stools (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (5) | 2 (4) | 2 (2) | 1 (2) | 21 (41) | 25 (62) | 25 (59)
Odynophagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oral Pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pancreatitis Acute (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Paraesthesia Oral (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Periodontal Disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Proctalgia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 4 (6) | 3 (3)
Rectal Discharge (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rectal Haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 3 (5) | 2 (2)
Rectal Tenesmus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 8 (9) | 18 (37) | 21 (35)
Subileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tongue Ulceration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tooth Discolouration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tooth Disorder (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (3) | 1 (1) | 2 (6) | 14 (21) | 12 (24) | 17 (30)
Asthenia (General disorders) | 0 (0) | 1 (2) | 3 (3) | 1 (1) | 9 (15) | 15 (26) | 20 (66)
Catheter Site Erythema (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Catheter Site Rash (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chest Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Chills (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 3 (4)
Extravasation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 15 (21) | 16 (26) | 17 (33)
Feeling Cold (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
General Physical Health Deterioration (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Impaired Healing (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Influenza Like Illness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (2)
Injection Site Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Localised Oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Malaise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mucosal Inflammation (General disorders) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Non-Cardiac Chest Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Oedema Peripheral (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (4) | 4 (5) | 3 (5)
Performance Status Decreased (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 4 (5) | 13 (23) | 8 (19)
Secretion Discharge (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Xerosis (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Biliary Colic (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cholestasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hepatic Pain (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hepatic Vein Thrombosis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hepatomegaly (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 4 (16) | 3 (4)
Jaundice (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 1 (1)
Contrast Media Allergy (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Drug Hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Abdominal Wall Abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anal Abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 4 (5) | 0 (0)
Catheter Site Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (3)
Cystitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 3 (7) | 2 (4)
Device Related Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Escherichia Urinary Tract Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eye Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Folliculitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Fungal Skin Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Furuncle (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 1 (1) | 0 (0)
Gastroenteritis Viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Genital Candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Herpes Zoster (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (3) | 0 (0)
Hordeolum (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Infected Fistula (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Infected Skin Ulcer (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (5) | 0 (0) | 2 (2)
Keratitis Herpetic (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Laryngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Localised Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lower Respiratory Tract Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lung Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lyme Disease (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nail Bed Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 5 (5) | 2 (2) | 4 (4)
Oesophageal Candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oral Candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 5 (5)
Oral Fungal Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4)
Oral Herpes (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (3)
Oral Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Otitis Externa (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Paronychia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 11 (25) | 6 (10) | 5 (9)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pharyngotonsillitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Postoperative Wound Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pulpitis Dental (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash Pustular (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (5) | 1 (1) | 0 (0)
Rhinitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 6 (7) | 3 (4)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Severe Acute Respiratory Syndrome (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (2) | 1 (1)
Streptococcal Urinary Tract Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Subcutaneous Abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tinea Pedis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tonsillitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Upper Respiratory Tract Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 6 (7) | 3 (4) | 4 (4)
Urinary Tract Infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 3 (7) | 6 (8) | 6 (7)
Viral Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (3)
Viral Upper Respiratory Tract Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vulvovaginal Mycotic Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Contrast Media Reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Head Injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Incisional Hernia (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Infusion Related Reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 4 (5) | 1 (1)
Post Procedural Discharge (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Post Procedural Haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Procedural Pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Radius Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sunburn (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Suture Related Complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wound (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Activated Partial Thromboplastin Time (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Activated Partial Thromboplastin Time Prolonged (Investigations) | 1 (5) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 4 (4) | 0 (0)
Alanine Aminotransferase Increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 12 (22) | 4 (5) | 3 (5)
Aspartate Aminotransferase Increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 8 (9) | 4 (4) | 4 (7)
Blood Alkaline Phosphatase Increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 4 (7) | 2 (3) | 6 (10)
Blood Bilirubin Increased (Investigations) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 2 (4)
Blood Glucose Increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (12)
Blood Iron Decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood Lactate Dehydrogenase Increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (10) | 1 (1)
Blood Magnesium Decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood Pressure Increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Blood Thyroid Stimulating Hormone Decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Blood Thyroid Stimulating Hormone Increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 0 (0)
Body Temperature Increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 1 (1) | 0 (0) | 0 (0)
C-Reactive Protein Increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Creatinine Renal Clearance Decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ejection Fraction Decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Electrocardiogram T Wave Inversion (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Eosinophil Count Increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gamma-Glutamyltransferase Increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (10) | 1 (1) | 3 (6)
Haematocrit Decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemoglobin Decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 1 (1)
International Normalised Ratio Increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 3 (4) | 0 (0)
Neutrophil Count Decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 0 (0) | 3 (6)
Neutrophil Count Increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Platelet Count Increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Red Blood Cell Count Decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thrombin Time Prolonged (Investigations) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Transaminases Increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urine Output Decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Weight Decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 7 (7) | 10 (12)
Weight Increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
White Blood Cell Count Increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cachexia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Decreased Appetite (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 3 (3) | 0 (0) | 9 (11) | 11 (15) | 20 (36)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 3 (3) | 3 (3)
Diabetes Mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (4) | 2 (5) | 2 (5)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypermagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 3 (4) | 2 (2)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 5 (6) | 11 (29) | 8 (12)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (5) | 4 (4) | 13 (27) | 15 (27)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (5) | 1 (1) | 1 (1) | 2 (5) | 17 (38) | 23 (57) | 14 (40)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (4) | 2 (3) | 3 (4)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (4) | 1 (1) | 9 (19)
Hypoproteinaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Iron Deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Malnutrition (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Plasma Protein Metabolism Disorder (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Type 2 Diabetes Mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (7) | 3 (3) | 2 (2)
Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 5 (5) | 3 (5) | 9 (10)
Flank Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Groin Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Inguinal Mass (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Joint Swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Mobility Decreased (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 2 (3) | 4 (5)
Muscle Twitching (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 0 (0) | 2 (2)
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Osteopenia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 4 (8)
Soft Tissue Disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Synovitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Cholinergic Syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 3 (4) | 2 (3) | 2 (3)
Diabetic Neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (4) | 1 (1)
Dizziness Postural (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 8 (8)
Encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Epilepsy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (2) | 3 (3)
Hepatic Encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Hypogeusia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lethargy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (6) | 2 (3) | 3 (4)
Neuropathy Peripheral (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neurotoxicity (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Peripheral Motor Neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Peripheral Sensory Neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (4) | 0 (0) | 2 (2)
Polyneuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 2 (2) | 1 (1)
Radiculitis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Sciatica (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Speech Disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Toxic Neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Visual Field Defect (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Agitation (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (4) | 1 (1) | 0 (0)
Confusional State (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Decreased Interest (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Depressed Mood (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Depressive Symptom (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Emotional Disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 4 (6)
Anuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 4 (5) | 2 (3)
Glycosuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 2 (3)
Leukocyturia (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Oliguria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Polyuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Proteinuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (5)
Renal Colic (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Renal Pain (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urethral Obstruction (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary Retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Balanitis (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Breast Mass (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Breast Pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haematospermia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pelvic Pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vulvovaginal Pruritus (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Asthmatic Crisis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bronchial Secretion Retention (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 7 (8) | 6 (6) | 3 (3)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 2 (2)
Dyspnoea Exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 4 (5) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (4) | 0 (0) | 0 (0) | 1 (2) | 7 (8) | 5 (6) | 7 (8)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Nasal Dryness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Obstructive Airways Disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (6)
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pulmonary Toxicity (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory Disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 0 (0)
Rhinitis Allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sputum Discoloured (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Throat Irritation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (6) | 0 (0) | 12 (26) | 7 (18) | 12 (33)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (2) | 2 (2) | 19 (26) | 12 (19) | 15 (26)
Dermal Cyst (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Dermatitis Acneiform (Skin and subcutaneous tissue disorders) | 1 (3) | 0 (0) | 3 (7) | 1 (5) | 13 (19) | 14 (41) | 18 (42)
Dermatitis Allergic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dermatitis Atopic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (5) | 0 (0)
Drug Eruption (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (6) | 0 (0) | 4 (5)
Dry Skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 9 (14) | 9 (19) | 11 (16)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (3) | 1 (1) | 2 (2) | 5 (14) | 2 (4)
Exfoliative Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hypertrichosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (4)
Ingrowing Nail (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 1 (2)
Intertrigo (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nail Disorder (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (2) | 0 (0)
Nail Toxicity (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (4)
Night Sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Onychoclasis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Palmar-Plantar Erythrodysaesthesia Syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 7 (10) | 7 (12) | 7 (16)
Panniculitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Penile Ulceration (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Petechiae (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pigmentation Disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Prurigo (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 6 (8) | 9 (13) | 10 (15)
Pruritus Generalised (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (4) | 3 (5) | 1 (3) | 3 (4) | 37 (75) | 37 (103) | 28 (76)
Rash Generalised (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (4)
Rash Papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 3 (4) | 1 (6)
Rash Pruritic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (6)
Rash Vesicular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin Chapped (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin Erosion (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin Exfoliation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Skin Fissures (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 9 (12) | 5 (14) | 5 (8)
Skin Irritation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Skin Ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2)
Subcutaneous Nodule (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Toxic Skin Eruption (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 1 (5) | 2 (5)
Aortic Thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Circulatory Collapse (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Deep Vein Thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 2 (3)
Flushing (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Haematoma (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 2 (2) | 3 (3)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (3) | 5 (6)
Orthostatic Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pallor (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Peripheral Ischaemia (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Phlebitis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Thrombophlebitis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Venous Insufficiency (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Venous Thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other